CLINICAL TRIAL: NCT07342829
Title: Prospective On-site Study for the Immunological Follow-up of Individuals Who Received Booster Vaccination With MVA-BN Against Mpox
Brief Title: Prospective Follow-up After MVA-BN Booster Vaccination
Acronym: POQS-Boosted
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: POQS-Boosted
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Monkeypox (Mpox)
Keywords: mpox; immunology; vaccination; booster
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum; Saliva; Anorectal swabs; PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
POQS-Boosted is a prospective observational study during which individuals who received Booster vaccination against mpox with the MVA-BN vaccine will be invited to provide biological samples at multiple times over the course of two years.

DETAILED DESCRIPTION:
Mpox caused a worldwide outbreak in 2022 and continues to circulate worldwide and causes sporadic cases in Belgium and elsewhere. In the last 10 days, the first cases infected with the probably more virulent clade Ib MPXV have been reported from men who have sex with men in Belgium, the Netherlands, and elsewhere, indicating circulating this viral clade in sexual networks. In Belgium, vaccination against mpox was ceased at the end of 2022 and evidence showed that antibody levels against MPXV have decreased since then, raising questions about sustained protectiveness and the potential for a new mpox outbreak to emerge.

POQS-Boosted is a prospective observational study during which individuals who received Booster vaccination against mpox with the MVA-BN vaccine will be invited to provide biological samples at multiple times over the course of two years.

ELIGIBILITY:
Inclusion Criteria:

1. Is scheduled to receive a booster dose of MVA-BN
2. ≥18 years
3. Willingness to provide written informed consent
4. Willingness to follow the study schedule

Exclusion Criteria:

1. Past or current MPXV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who received MVA-BN booster vaccination will be asked to participate in "POQS-Boosted"
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Orthopoxvirus-specific serum binding and neutralising antibody titre | from enrollment to the end of follow up at 2 years
  To describe the evolution of the orthopoxvirus-specific serum antibody response up to two years after MVA-BN booster vaccination

SECONDARY OUTCOMES:
Orthopoxvirus-specific systemic T- and B cell-mediated immune responses to MPXV | from enrollment up to 2 years
  To describe the evolution of the orthopoxvirus-specific systemic cellular immune response up to two years after MVA-BN booster vaccination
MPXV-specific IgA in saliva and anorectal samples; T and B cell-mediated immune responses to MPXV, measured on saliva and anorectal samples | from enrolment up to two years
  To describe the evolution of the orthopoxvirus-specific mucosal antibody & cellular immune response up to two years after MVA-BN booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, MD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided